CLINICAL TRIAL: NCT04815252
Title: Testing the Initial Efficacy of a Mindfulness Compassion-based Intervention to Support Wellbeing Amongst Early Childhood Professionals
Brief Title: Mindfulness Intervention for Early Childhood Educators
Acronym: CHIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20336
Record Dates: First submitted 2020-08-27; First posted 2021-03-24 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Stress, Psychological; Stress, Physiological
Keywords: Mindfulness; Early childhood educator; Intervention; Burnout
MeSH Terms: conditions — Stress, Psychological; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Participants are assigned, based on childcare center, to the intervention or waitlist control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHIME Intervention (Experimental): Participants will complete an 8-week compassion and mindfulness-based intervention with a group facilitator. The curriculum focuses on providing mindfulness-based stress reduction techniques for use in the early childhood education environment.
  Interventions: Behavioral: CHIME
- Waitlist control (No Intervention): Participants are placed on a wait-list to receive the intervention.

INTERVENTIONS:
Behavioral: CHIME — CHIME is a professional development program to provide knowledge and skills for nurturing early childhood educator mindfulness, compassion and socio-emotional learning. CHIME is a manualized curriculum delivered by a trained facilitator. The intervention consists of a 2-hour overview and seven weekly sessions, each lasting 90 minutes. Sessions can be delivered online or in-person.
  Arms: CHIME Intervention

SUMMARY:
This is a randomized trial of the 'Cultivating Healthy, intentional, Mindful Educators' (CHIME) intervention designed for early childhood educators. The intervention aims to enhance wellbeing, emotion regulation, and sensitive, responsive caregiving among educators by providing them with mindfulness, compassion-based techniques to alleviate stress and respond to emotional challenges in the classroom. The intervention ultimately aims to enhance children's self-regulation through sensitive, responsive caregiving. Measures of teachers' emotional regulation, wellbeing, and stress physiology will be collected pre- and post- the 8 week intervention and compared to a waitlist comparison group. Measures of child self-regulation also will be collected to assess the relation of teacher stress, wellbeing and emotion regulation to child self-regulation.

DETAILED DESCRIPTION:
Across varied disciplines, the science is clear that early relationships and the quality of early care are central in achieving positive language, cognitive, and social development outcomes for young children and investments made in early childhood pay for themselves. Early childhood education is a critical context for fostering stimulating, responsive, and sensitive caregiving as a substantial number of children under the age of 5 years spend time in childcare settings, with 64% of children aged 3 to 5 years enrolled in non-relative care outside the home. While great efforts are made to improve the children's social emotional well-being in child care environments, less attention has been given to early childhood educators' (encompassing of early childhood teachers') own well-being. Research that has been conducted finds early childhood educators experience high levels of distress, including high levels of depression and burnout. Additionally, previous research finds school age teachers feeling overworked and overstressed show an altered hypothalamus-pituitary-adrenal (HPA) axis and higher levels of teacher burnout is related to elevated cortisol levels in elementary school students.

The current study will test the efficacy of an 8-week compassion and mindfulness based stress reduction program for early childhood educators, as well as characterizing relations from early childhood educator wellbeing to child self-regulation. Teachers will be assigned at the center level to an intervention group or a wait-list comparison condition, with the wait-list group receiving the intervention after the 8-week study. Pre- intervention, teachers in both groups will complete survey measures of their wellbeing, mindfulness, and emotion regulation; emotion regulation tasks; and assessments of stress physiology in the classroom. Teacher-child interactions will be observed and children's self-regulation will be measured. Post-intervention, the same teacher measures will be collected.

ELIGIBILITY:
Inclusion Criteria:

Teachers/educators:

* Providing care to children aged birth through 6 years
* Participating in, or are signed up to eventually participate in, the 8-week "Cultivating Healthy Intentional, Mindful Educators" (CHIME) intervention
* English speakers
* 19 years of age or older.

Children:

* Aged 3-6 years
* Enrolled in a preschool setting with a teachers enrolled/signed up to participate in the CHIME study.
* English or Spanish speakers

Parents:

* Have a child aged 3-6 who is enrolled in a preschool classroom of a teacher participating in the study.
* Speak and read English or Spanish and
* Legal guardian
* 19 years of age or older.

Exclusion Criteria:

*Not participating/enrolled to participate in CHIME

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change on the Cognitive and Affective Mindfulness Scale Revised | Week 1, week 9
  Measures attention regulation, awareness, acceptance, and mindful focus on the present. The scale comprises 12 items rated on a 5-point scale. Scores on this scale range from 12-60, with higher scores indicating greater levels of mindfulness.
Change on the Self Compassion Scale - Short Form | Week 1, Week 9
  Measures the tendency to treat oneself with compassion, mindfulness and feelings of isolation. The scale comprises 12 items, with scores ranging from 12-60. Higher scores indicate greater levels of self-compassion.
Change on the Emotion Regulation Questionnaire | Week 1, Week 9
  Measures the tendency to engage in cognitive reappraisal or suppression of negative emotions. The reappraisal scale comprises 6 items with scores ranging from 6-42. the suppression scale comprises 4 items with scores ranging from 4-28. Higher levels of reappraisal and lower levels of suppression are associated with better emotion regulation.
Change on the Difficulties in Emotion Regulation Scale | Week 1, Week 9
  Measures emotional awareness, clarity and strategy use, and impulse control. The scale comprises 36 items rated on a 5-point scale, with total scores ranging from 36-180. Higher scores indicate higher levels of difficulty regulating emotions.
Change on the Emotion Stroop | Week 1, Week 9
  Computerized task administered online that measures the ability to override attentional interference from emotion. A greater difference in the reaction times for emotional vs. neutral trials indicates greater in difficulty in over-riding attentional interference from emotion.
Change on the Modified Emotional Exogenous Cuing Paradigm | Week 1, Week 9
  Computerized task administered online that measures the ability to override attentional interference from emotion. Longer reaction times during incongruent emotional trials relative to neutral emotional trials indicate greater difficulty resisting attentional interference from emotion.
Change on the Short Warwick-Edinburgh Mental Wellbeing Measure | Week 1, Week 9
  A Rasch-validated questionnaire that captures feelings of happiness, social wellbeing and quality of life. Scores range from 14-70, with higher scores indicating higher levels of wellbeing.
Change on the The Early Childhood Job Attitude Survey | Week 1, week 9
  A questionnaire that evaluates workplace satisfaction and supports and workload manageability. Scores range from 5-25, with higher scores indicating more negative workplace perceptions.
Change on the Job Demands scale | Week 1, week 9
  Taken from the Child Care Worker Job Stress Inventory, this questionnaire will provide a more detailed assessment of stress related to parent interactions and challenging child behavior. The scale comprises 16 items rated on a scale from 1-5. Total scores range from 16-80, with higher scores indicative of greater stress.
Change on the The Effort/Reward imbalance scale | Week 1, week 9
  This questionnaire measures the balance of effort relative to reward that people feel they are putting into their work. The effort-reward imbalance ratio is calculated as the effort score, which ranges from 5-25, divided by the reward score (ranging from 11-55) multiplied by a correction factor. The minimum score is 0 and values above 1 are less favorable and indicate a high level of effort relative to workplace reward.
Change in Salivary Cortisol | Week 1, week 9
  Measure of the reactivity of the hypothalamic pituitary-adrenal axis. Saliva will be collected by passive drool in the morning and in the afternoon for two consecutive days.
Change in the Heart rate variability | Week 1, Week 9
  Teachers will wear an 'Actiheart' device to measure cardiac inter-beat intervals and motion for three consecutive days in the classroom. Root mean square of successive differences will be calculated as a measure of heart rate variability.
Change in Classroom Assessment Scoring System Emotional Support score | Week 1, week 9
  Teacher behavior will be observed and coded using the Emotional Support scale from the Classroom Assessment Scoring System. The primary outcome is the Emotional Support scale, which centers on the teachers' capacity to create a sensitive and positive emotional climate in the classroom. Scores range from 0 to 7, with scores of 7 indicating higher levels emotional support.

OTHER OUTCOMES:
Child self-regulation task | Week 1
  This measure will be administered through 'Zoom.' Children are instructed to respond to directions from one puppet, but to inhibit their behavioral responses to another puppet. Scores range from 0-100, with higher scores indicating higher levels of self-regulation.
Behavioral Rating Inventory of Executive Function - Preschool | Week 1
  This questionnaire measure will be completed by parent or legal guardians to assess children's self-regulation of emotion and behavior in everyday settings. The total score is rated on a t-score metric, with higher scores reflecting higher levels of difficulty in executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Caron Clark, Principal Investigator — UNL; Holly Hatton-Bowers, Principal Investigator — UNL
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Scored and de-identified data that is stripped of any information that could be used to identify participants may be shared. Data will not be shared if there is any possibility that participants or childcare centers may be identifiable (e.g., based on geographic region).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the data.
Access Criteria: Researchers may contact the study team to obtain information.

REFERENCES:
- [Background] Cassidy, D. J., Lippard, C., King, E. K., & Lower, J. K. (2019). Improving the Lives of Teachers in the Early Care and Education Field to Better Support Children and Families. Family Relations. https://doi.org/10.1111/fare.12362
- [Background] Curbow, B., Spratt, K., Ungaretti, A., McDonnell, K., & Breckler, S. (2000). Development of the child care worker job stress inventory. Early Childhood Research Quarterly, 15(4), 515-536. https://doi.org/10.1016/S0885-2006(01)00068-0
- [Background] Feldman, G., Hayes, A., Kumar, S., Greeson, J., & Laurenceau, J. (2007). Mindfulness and Emotion Regulation: The Development and Initial Validation of the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Journal of Psychopathology and Behavioral Assesssment, 29, 177-190. https://doi.org/10.1007/s10862-006-9035-8
- [Background] Flook L, Goldberg SB, Pinger L, Bonus K, Davidson RJ. Mindfulness for teachers: A pilot study to assess effects on stress, burnout and teaching efficacy. Mind Brain Educ. 2013 Sep;7(3):10.1111/mbe.12026. doi: 10.1111/mbe.12026. PMID 24324528
- [Background] Gioia, G. A., Espy, K. A., & Isquith, P. K. (2003). BRIEF-P: Behavior Rating Inventory of Executive Function - Preschool Version. Lutz, FL: Psychological Assessment Resources.
- [Background] Gotlib IH, McCann CD. Construct accessibility and depression: an examination of cognitive and affective factors. J Pers Soc Psychol. 1984 Aug;47(2):427-39. doi: 10.1037//0022-3514.47.2.427. PMID 6481620
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54. https://doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Howard SJ, Melhuish E. An Early Years Toolbox for Assessing Early Executive Function, Language, Self-Regulation, and Social Development: Validity, Reliability, and Preliminary Norms. J Psychoeduc Assess. 2017 Jun;35(3):255-275. doi: 10.1177/0734282916633009. Epub 2016 Feb 28. PMID 28503022
- [Background] Jeon, L., Buettner, C. K., Grant, A. A., Jeon, L., Buettner, C. K., & Early, A. A. G. (2018). Early Childhood Teachers' Psychological Well-Being: Exploring Potential Predictors of Depression , Stress , and Emotional Exhaustion Early Childhood Teachers ' Psychological Well-Being : Exploring. Early Education and Development, 29(1), 53-69. https://doi.org/10.1080/10409289.2017.1341806
- [Background] Mamedova, S., & Redford, J. (2015). Early childhood program participation, From the National Household Education Surveys Program of 2012. Washington D.C.
- [Background] McClelland, M. M., & Wanless, S. B. (2012). Growing up with assets and risks: The importance of self-regulation for academic achievement. Research in Human Development, 9(4), 278-297. https://doi.org/10.1080/15427609.2012.729907
- [Background] Neff, K. D. (2003). Measure - Self-Compassion Scale (SCS). Self and Identity, 2, 223-250. https://doi.org/10.1080/15298860309027
- [Background] Oberle E, Schonert-Reichl KA. Stress contagion in the classroom? The link between classroom teacher burnout and morning cortisol in elementary school students. Soc Sci Med. 2016 Jun;159:30-7. doi: 10.1016/j.socscimed.2016.04.031. Epub 2016 Apr 24. PMID 27156042
- [Background] Roberts, A., LoCasale-Crouch, J., Hamre, B., & DeCoster, J. (2016). Exploring Teachers' Depressive Symptoms, Interaction Quality, and Children's Social-Emotional Development in Head Start. Early Education and Development, 27(5), 642-654. https://doi.org/10.1080/10409289.2016.1127088
- [Background] Siegrist J, Starke D, Chandola T, Godin I, Marmot M, Niedhammer I, Peter R. The measurement of effort-reward imbalance at work: European comparisons. Soc Sci Med. 2004 Apr;58(8):1483-99. doi: 10.1016/S0277-9536(03)00351-4. PMID 14759692
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Carlson SM. Developmentally sensitive measures of executive function in preschool children. Dev Neuropsychol. 2005;28(2):595-616. doi: 10.1207/s15326942dn2802_3. PMID 16144429